CLINICAL TRIAL: NCT03816488
Title: Oral Peri-operative TIming of Metformin (or) Salsalate to Improve Non-cardiac Surgery Glucose Control - A Placebo-Controlled Internal Feasibility Trial
Brief Title: Oral Peri-operative TIming of Metformin (or) Salsalate to Improve Non-cardiac Surgery Glucose Control
Acronym: OPTIM(i)SING
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to source salsalate.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5451
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia; Perioperative/Postoperative Complications
Keywords: Metformin; Salsalate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Postoperative Complications | interventions — Metformin; salicylsalicylic acid

STUDY DESIGN:
Intervention Model Description: Parallel, placebo-controlled trial with block randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized on the day of their pre-operative assessment by our department statistician using a computer-generated table, with an allocation ratio of 1:1:1 in random permuted blocks of 3 or 6. Only the pharmacist and statistician will know the allocation sequence. Concealed medications (over-encapsulated) will be provided to the RC upon confirming the allotment with a unique identification number (UIN), recorded on the patient-specific case record form (CRF).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin (Experimental): Self-administered metformin (patient's usual dose) taken 2 hours prior to surgery
  Interventions: Drug: Metformin
- Salsalate (Experimental): Self-administered salsalate taken 2 hours prior to surgery
  Interventions: Drug: Salsalate
- Placebo (No Intervention): Self-administered placebo taken 2 hours prior to surgery

INTERVENTIONS:
Drug: Metformin — Metformin (usual dose) administered 2 h before surgery
  Arms: Metformin
Drug: Salsalate — Salsalate 1.5 g administered 2 h before surgery
  Arms: Salsalate

SUMMARY:
Hypothesis: In surgical patients with type 2 diabetes, taking either metformin or salsalate on the morning of surgery will reduce the incidence of hyperglycemia, inflammation and even surgical site infections, without any obvious patient risk relative to patients given a placebo control.

Anesthesia and surgery induce a number of metabolic disturbances, particularly among patients with type 2 diabetes (T2D). This includes altered glucose metabolism and hyperglycemia, which is associated with significant morbidity and mortality, including an increase in surgical site infections (SSI). Although insulin protocols can reduce blood glucose levels in hyperglycemic surgical patients, leading to reduced SSI, this has caused severe hypoglycemia in a number of patients. Instead, the use of simple and effective interventions, such as continuing metformin on the day of surgery, could represent an important step toward reducing the incidence of these morbid outcomes while improving glucose control. Alternatively, salsalate, a non-acetylated dimer of salicylic acid, has also emerged as a novel glucose-lowering medication that also possesses important anti-pyretic and anti-inflammatory properties and could prove equally effective.These refinements may also reduce SSI and inflammation. If the proposed pilot trial, to continue metformin, or take salsalate, peri-operatively, is as safe and easy as the investigators anticipate it will allow for the planning of a future definitive randomized clinical trial. The aims of this pilot trial are to assess the feasibility of safely continuing metformin, or taking salsalate on the day of surgery, with the goal of reducing the incidence of hyperglycemic events. This includes assessing our ability to recruit patients, adhere to the proposed study protocol, assess workload,and measure the desired outcomes, all of which are crucial for the planning of a subsequent clinical trial.

DETAILED DESCRIPTION:
This internal pilot study (n=36) is designed as a 3-arm, parallel, placebo-controlled trial with block randomization. All parties will be blinded.

Patient Recruitment: Patients with T2D on metformin presenting to the Hamilton Health Sciences (HHS) preoperative clinic for elective surgery requiring general anesthetic will be screened for eligibility.

Sample Size: 36 patients over the 1-year study. This sample size will allow for 3 groups of 12, which permits block randomization and precise confidence interval (CI) calculations.

Randomization and Allocation: Patients will be randomized on the day of their pre-operative assessment by our department statistician using a computer-generated table, with an allocation ratio of 1:1:1 in random permuted blocks of 3 or 6. Only the pharmacist and statistician will know the allocation sequence. Concealed medications (over-encapsulated) will be provided to the RC upon confirming the allotment with a unique identification number (UIN), recorded on the patient-specific case record form (CRF).

Application of Intervention: Our intervention involves self-administered metformin (patient's usual dose) vs. salsalate (1.5g) vs. placebo with sips of water 2h prior to surgery. Baseline data (age, height, weight, ASA score, mean arterial BP, and baseline glucose) will be collected by the RC in the pre-operative assessment area, and flash glucose sensors (FreeStyle Libre, Abbot) will be placed on the upper arm as per manufacturer's instructions and readings collected by the RC. Study data will be securely stored in the anesthesia research office, McMaster University. Standard monitors will be used in the operating room, with any additional monitoring left to the anesthesiologist's discretion. Although most anesthetics appear to modify glucose metabolism, general anesthesia will be provided in their preferred manner (including dexamethasone administration for post-operative nausea and vomiting prophylaxis) to improve generalizability. Details of the type of drugs, fluids and blood loss will be recorded. Following surgery, patients will be brought to the PACU for routine monitoring (30-60 min), and additional blood samples will be drawn. Subsequent samples will be collected on the evening of surgery (6-12h) and POD1. Any episodes of hyper- or hypoglycemia will be managed routinely at the treating physician's discretion and details recorded.

Measurements of Inflammation: Blood and urine samples will be collected on the morning of surgery, upon admission to PACU, and will coincide with other tests to minimize needle sticks. Blood samples will be processed at the HHS Core Research Laboratory and divided into 3 serum and 2 EDTA aliquots, barcoded and stored in liquid nitrogen. Urine samples will be divided into 2 barcoded aliquots and stored in liquid nitrogen. This will allow for future analysis and characterization of biochemical pathways related to the surgical stress response. These future analyses will include measurement of insulin and proinsulin since salsalate may modify their endogenous metabolism. Similarly, the investigators eventually plan to measure various inflammatory markers implicated in the development of acute stress-induced insulin resistance (i.e. IL-6, TNFα, and hsCRP), which could provide insight into potential beneficial effects of salsalate or metformin.

Feasibility Outcomes: The primary feasibility outcomes include calculating the recruitment rate (both the percentage of individuals who were approached in the pre-operative clinic that enrolled in the study, and the total number of individuals that were recruited each month (Table 1, supplemental document). The ability to follow study protocol will be reported as the percentage of individuals who were able to complete the study protocol as a fraction of the total number of individuals recruited for i) drug administration and blinding, ii) blood sampling at specified times, and iii) reliability of CGM by comparison with laboratory glucose values. Workload will be calculated per patient, and safety profile assessed by recording adverse events. Together, this may identify pitfalls requiring modification prior to a full RCT.

Statistical Analysis and Feasibility: Reporting and analysis will conform to the CONSORT pilot and feasibility trials guidelines (www.consort-statement.org). Data will be collected using an encrypted online tool (RedCap, Research Electronic Data Capture) hosted at McMaster. To be feasible and continue onto a subsequent RCT the investigators will need to recruit at least 3 patients per month. Additionally, the investigators seek an adherence rate of 88.9% (32/36) to receive study drug, collect more than 90.3% (130/144) of pre-specified blood samples, and ensure 83.3% (30/36) patients have been followed up within 6 weeks of their procedure to document any complications (e.g. SSI). If targets prove difficult, then our protocol will be reevaluated for possible amendments that will not compromise final outcomes. Given this is a pilot, CIs will be calculated for outcomes of interest: rates of hyperglycemia, SSI, and degree of inflammation.

Trial Management: This pilot trial will be conducted at HHS. The trial will enlist support and collaboration from surgeons and fellow anesthesiologists. Study data will be securely stored at the anesthesia research office, McMaster University. An RC will be employed for patient recruitment and data collection. The CRFs for study patients will be randomly cross-checked for completeness and accuracy. All reports of incorrect randomizations, protocol violations or incomplete data will be noted.

Risk Assessment: This trial does not entail any higher risk to the patient than the present standard of care. It is pragmatic, and uses clinically acceptable doses with a safe profile.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients requiring a general anesthetic at HHS requiring at least an overnight admission;
* Using metformin regularly for control of T2D;
* American Society of Anesthesiologists (ASA) physical classification I, II and III;
* Less than 1000 mL of blood loss is expected.

Exclusion Criteria:

* Procedures for which non-steroidal anti-inflammatory drugs are contraindicated;
* Diagnosis of renal failure (estimated glomerular filtration rate <60 mL/min/1.73m2);
* Liver failure;
* Previous episodes of congestive heart failure;
* Severe hypoglycemia in the past year;
* Conditions masking hypoglycemia (e.g. autonomic neuropathy);
* Low random blood glucose during pre-screening (≤4.0 mmol/L);
* Received contrast within 48h prior to, or during, surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: recruitment rate (percentage) | One year
  Percentage (%) of individuals who were approached in the pre-operative clinic that enrolled in the study
Participants with hyperglycemia | One year
  Detect change in hyperglycemic events (glucose >11mmol/L) at the 4 blood sampling time points for each participant
Feasibility: recruitment rate (total number per month) | One year
  Number (n) of individuals recruited each month

SECONDARY OUTCOMES:
Blood glucose levels (glycemic control) | One year
  Evaluation of glycemic control by calculating mean blood glucose levels obtained at 4 time points
Number of participants with inflammation | One year
  Measured using validated biomarkers (IL-6, tumor necrosis factor, high-sensitivity C reactive protein), and surgical site infections recorded within 6 weeks of surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palermo NE, Gianchandani RY, McDonnell ME, Alexanian SM. Stress Hyperglycemia During Surgery and Anesthesia: Pathogenesis and Clinical Implications. Curr Diab Rep. 2016 Mar;16(3):33. doi: 10.1007/s11892-016-0721-y. PMID 26957107
- [Background] Frisch A, Chandra P, Smiley D, Peng L, Rizzo M, Gatcliffe C, Hudson M, Mendoza J, Johnson R, Lin E, Umpierrez GE. Prevalence and clinical outcome of hyperglycemia in the perioperative period in noncardiac surgery. Diabetes Care. 2010 Aug;33(8):1783-8. doi: 10.2337/dc10-0304. Epub 2010 Apr 30. PMID 20435798
- [Background] Membership of the Working Party; Barker P, Creasey PE, Dhatariya K, Levy N, Lipp A, Nathanson MH, Penfold N, Watson B, Woodcock T. Peri-operative management of the surgical patient with diabetes 2015: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2015 Dec;70(12):1427-40. doi: 10.1111/anae.13233. Epub 2015 Sep 29. PMID 26417892
- [Background] Smith BK, Ford RJ, Desjardins EM, Green AE, Hughes MC, Houde VP, Day EA, Marcinko K, Crane JD, Mottillo EP, Perry CG, Kemp BE, Tarnopolsky MA, Steinberg GR. Salsalate (Salicylate) Uncouples Mitochondria, Improves Glucose Homeostasis, and Reduces Liver Lipids Independent of AMPK-beta1. Diabetes. 2016 Nov;65(11):3352-3361. doi: 10.2337/db16-0564. Epub 2016 Aug 23. PMID 27554471